CLINICAL TRIAL: NCT04715113
Title: Hemodynamic Effects of Acute Normobaric Hypoxia During Exercise in Patients With Pulmonary Hypertension: Single-center Randomized Controlled Trial
Brief Title: Blood Markers Predict Effect of Normobaric Hypoxia at Rest and During Exercise in Patients With Pulmonary Hypertension
Acronym: HEXABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-02163_A4
Record Dates: First submitted 2020-12-20; First posted 2021-01-20 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Pulmonary
Keywords: hypoxia; exercise; blood markers
MeSH Terms: conditions — Hypertension, Pulmonary; Hypoxia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normobaric hypoxia (FiO2 15%) (Experimental): Inhalation of deoxygenated air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Interventions: Other: Normobaric hypoxia (FiO2 15%)
- Placebo-ambient air (FiO2 21%) (Sham Comparator): Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Interventions: Other: Placebo-ambient air (FiO2 21%)
- Normobaric hypoxia (FiO2 15%) under Sildenafil (Experimental): Inhalation of deoxygenated air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Interventions: Other: Normobaric hypoxia (FiO2 15%) under Sildenafil
- Placebo-ambient air (FiO2 21%) under Sildenafil (Active Comparator): Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Interventions: Other: Placebo-ambient air (FiO2 21%) under Sildenafil

INTERVENTIONS:
Other: Normobaric hypoxia (FiO2 15%) — Inhalation of deoxygenated air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Arms: Normobaric hypoxia (FiO2 15%)
Other: Placebo-ambient air (FiO2 21%) — Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Arms: Placebo-ambient air (FiO2 21%)
Other: Normobaric hypoxia (FiO2 15%) under Sildenafil — Inhalation of deoxygenated air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise under Sildenafil.
  Arms: Normobaric hypoxia (FiO2 15%) under Sildenafil
Other: Placebo-ambient air (FiO2 21%) under Sildenafil — Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise under Sildenafil.
  Arms: Placebo-ambient air (FiO2 21%) under Sildenafil

SUMMARY:
To study the effect of acute normobaric hypoxia during exercise in patients with pulmonary hypertension on blood markers (serum markers of iron and red blood cell homeostasis and micro-RNAs known to be associated with PH).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zürich altitude on ambient air
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* patients who take nitrates
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Serum levels of ferritin | Baseline
  Analyis of serum levels of ferritin

SECONDARY OUTCOMES:
Serum levels of transferrin | Baseline
  Analyis of serum levels of transferrin
Serum levels of total iron | Baseline
  Analysis of serum levels of total iron
Serum levels of erythropoietin | Baseline
  Analysis of serum levels of erythropoietin
Serum levels of Erythroferrone | Baseline
  Analysis of serum levels of erythroferrone
Serum levels of hepcidin | Baseline
  Analysis of serum levels of hepcidin
micro-RNA levels | Baseline
  Analysis of micro-RNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — UniversityHospital Zurich, Department of Pulmonology
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data after publication of the manuscript. The decision about the platform is ongoing.
Time Frame: After publication of the manuscript